CLINICAL TRIAL: NCT00003181
Title: A Phase II Study Using Low Dose Subcutaneous IL-2, Vinblastine and GM-CSF in the Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Interleukin-2, Vinblastine, and GM-CSF in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hope Cancer Institute, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066003; HCRN-002; NCI-V98-1373
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-05

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; sargramostim; Vinblastine

INTERVENTIONS:
Biological: aldesleukin
Biological: sargramostim
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining chemotherapy with interleukin-2 and GM-CSF may be a more effective treatment for kidney cancer.

PURPOSE: Phase II trial to study the effectiveness of low-dose interleukin-2, vinblastine, and GM-CSF in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of sargramostim (granulocyte-macrophage colony-stimulating factor; GM-CSF) in combination with interleukin-2 and vinblastine on the response rate of patients with metastatic renal cell carcinoma. II. Assess the potential toxicities of this treatment combination in these patients.

OUTLINE: This is a single arm, nonrandomized study. Patients receive vinblastine as an IV bolus once every 2 weeks. Interleukin-2 is administered by subcutaneous injection on days 1-5 each week for 9 weeks. Sargramostim (granulocyte-macrophage colony-stimulating factor; GM-CSF) is administered by subcutaneous injection on days 1-5 each week for 9 weeks. Each 9 week cycle is followed by 3 weeks of rest. Patient may continue treatment for a maximum of 5 cycles in the absence of disease progression. Patients are assessed every 12 weeks for the duration of treatment.

PROJECTED ACCRUAL: 20-35 patients will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven inoperable, metastatic, or recurrent renal cell carcinoma Measurable or evaluable disease No brain metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: SWOG 0-2 Life expectancy: At least 3 months Hematopoietic: Neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Liver enzymes less than 3 (5 if known liver metastases) times institutional normal Renal: Creatinine less than 1.5 mg/dL Cardiovascular: Adequate cardiac function No unstable angina No significant coronary artery disease No heart failure with New York Heart Association classification III or IV Pulmonary: No evidence of pulmonary disease (documented normal DLCO and PFT) Other: No prior malignancy except: Nonmelanoma skin cancer Carcinoma in situ of any kind No pregnant or lactating Fertile patients must use adequate contraception Normal thyroid functions as evidenced by normal T4 and TSH

PRIOR CONCURRENT THERAPY: Biologic therapy: No more than 1 prior biologic therapy At least 4 weeks since prior biologic therapy Chemotherapy: No more than 1 prior chemotherapy At least 4 weeks since prior chemotherapy Endocrine therapy: No more than 1 prior hormonal therapy At least 4 weeks since prior hormonal therapy Radiotherapy: At least 4 weeks since prior radiation therapy No prior radiation therapy if entire tumor was within radiation field Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1997-05

CONTACTS AND LOCATIONS:
Overall Officials: Raj Sadasivan, MD, PhD, Study Chair — Hope Cancer Institute, Inc.
Locations (2):
- United States (2):
  - Bethany Medical Center, Kansas City, Kansas
  - Heartland Cancer Research and Treatment Center, Kansas City, Kansas